CLINICAL TRIAL: NCT04851964
Title: A Multicentre, Randomised, Double-Blind, Parallel-Group, Placebo-Controlled Phase 3 Efficacy and Safety Study of Tezepelumab in Participants With Severe Chronic Rhinosinusitis With Nasal Polyposis (WAYPOINT)
Brief Title: Efficacy and Safety of Tezepelumab in Participants With Severe Chronic Rhinosinusitis With Nasal Polyposis
Acronym: WAYPOINT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5242C00001; 2020-003062-39 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-04-21 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: Chronic rhinosinusitis with nasal polyps; Nasal polyps; Nasal polyposis
MeSH Terms: conditions — Nasal Polyps | interventions — Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either tezepelumab or matching placebo both administered subcutaneously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection in an accessorized pre-filled syringe every 4 weeks (Q4W) added to background mometasone furoate (MFNS) or equivalent intranasal corticosteroid (INCS).
  Interventions: Biological: Experimental: Tezepelumab; Drug: Mometasone furoate or equivalent intranasal corticosteroid
- Placebo (Placebo Comparator): Placebo subcutaneous injection in an accessorized pre-filled syringe Q4W added to background MFNS or equivalent INCS.
  Interventions: Other: Placebo; Drug: Mometasone furoate or equivalent intranasal corticosteroid

INTERVENTIONS:
Biological: Experimental: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo
Drug: Mometasone furoate or equivalent intranasal corticosteroid — Background MFNS or equivalent INCS at stable dose

SUMMARY:
A Multicentre, Randomised, Double-Blind, Parallel-Group, Placebo-Controlled Phase 3 Efficacy and Safety Study of Tezepelumab in Participants with Severe Chronic Rhinosinusitis with Nasal Polyposis

DETAILED DESCRIPTION:
This is a multicentre, randomised, double-blind, placebo controlled, parallel group study designed to evaluate the efficacy and safety of tezepelumab in adults with severe, chronic rhinosinusitis with nasal polyposis. Approximately 400 subjects will be randomized globally. Participants will receive tezepelumab, or placebo, administered via subcutaneous injection using the accessorized pre-filled syringe (APFS) every 4 weeks, over a 52-week treatment period. The study also includes a post-treatment follow-up period of 12-24 weeks for participants who complete the 52-week treatment period. All participants will have background mometasone furoate nasal spray or equivalent intranasal corticosteroid at a stable dose from Visit 1 and throughout the screening and study period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with physician-diagnosed CRSwNP for at least 12 months prior to Visit 1 that have:

   1. Severity consistent with need for surgery as defined by total NPS ≥ 5 (≥ 2 for each nostril) at screening, as determined by the central reader
   2. Nasal Congestion Score (NCS) ≥ 2 at Visit 1
   3. Ongoing documented NP symptoms over > 8 weeks prior to screening such as rhinorrhea and/or reduction/loss of smell
2. SNOT-22 total score ≥ 30 at screening (Visit 1)
3. Any standard of care for treatment of CRSwNP provided the participant is stable on that treatment for 30 days prior to Visit 1
4. Documented treatment of nasal polyposis exacerbation with SCS for at least 3 consecutive days or one IM depo-injectable dose (or contraindications/intolerance to) within the past 12 months prior to Visit 1 but not within the last 3 months prior to Visit 1 and/or any history of NP surgery (or contraindications/intolerance to)

Exclusion Criteria:

1. Any clinically important comorbidities other than asthma (e.g. active lung infection, bronchiectasis, pulmonary fibrosis, cystic fibrosis, primary ciliary dyskinesia, allergic bronchopulmonary mycosis, hypereosinophilic syndromes, etc.) that could confound interpretation of clinical efficacy results.
2. Sinus surgery within 6 months of screening visit OR any sinus surgery in the past which changed the lateral wall of the nose making NPS evaluation impossible.
3. Positive COVID-19 PCR test (or COVID-19 rapid test) or COVID-19 entry screening questionnaire during the screening visit. Evaluation will be based on on local standard of care as determined by current local guidelines.
4. Regular use of decongestants (topical or systematic) at enrolment is not allowed unless used for endoscopic procedure
5. Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, mycophenolate, tacrolimus, gold, penicillamine, sulfasalazine, hydroxychloroquine, systemic corticosteroids or any experimental anti-inflammatory therapy) within 3 months prior to Visit 1 and during the study period. Systemic corticosteroid use is defined as treatment with a burst of systemic corticosteroids for at least 3 consecutive days or a single IM depo-injectable dose of corticosteroids (considered equivalent to a 3-day burst of systemic corticosteroids).
6. Receipt of COVID-19 vaccine (regardless of vaccine delivery platform) 28 days prior to date of IP administration at Visit 3 (randomisation visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, MD, Principal Investigator — University of Dundee; Joseph K Han, MD, Principal Investigator — Eastern Virginia Medical School
Locations (100):
- United States (21):
  - Research Site, Birmingham, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Newport Beach, California
  - Research Site, Roseville, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Boca Raton, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Columbia, Missouri
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, North Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Milwaukee, Wisconsin
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- China (18):
  - Research Site, Bengbu
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hengyang
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
  - Research Site, Zunyi
- Denmark (8):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Køge
  - Research Site, Odense
  - Research Site, Vejle
- Germany (7):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Heidelberg
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Tübingen
  - Research Site, Wiesbaden
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Székesfehérvár
- Japan (18):
  - Research Site, Bunkyō City
  - Research Site, Chuo-shi
  - Research Site, Habikino-shi
  - Research Site, Ichikawa-shi
  - Research Site, Itabashi-ku
  - Research Site, Kashiwa-shi
  - Research Site, Kisarazu-shi
  - Research Site, Miyazaki
  - Research Site, Nagaoka-shi
  - Research Site, Nerima-ku
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Saitama-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Suwa-shi
  - Research Site, Toyonaka Shi
  - Research Site, Yokohama
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Nadarzyn
  - Research Site, Wroclaw
  - Research Site, Zawadzkie
  - Research Site, Łodź
- Spain (6):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Jerez de la Frontera
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- United Kingdom (4):
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Stockport

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Lipworth BJ, Han JK, Desrosiers M, Hopkins C, Lee SE, Mullol J, Pfaar O, Li T, Chen C, Almqvist G, Margolis MK, McLaren J, Jagadeesh S, MacKay J, Megally A, Hellqvist A, Mankad VS, Bahadori L, Ponnarambil SS; WAYPOINT Study Investigators. Tezepelumab in Adults with Severe Chronic Rhinosinusitis with Nasal Polyps. N Engl J Med. 2025 Mar 27;392(12):1178-1188. doi: 10.1056/NEJMoa2414482. Epub 2025 Mar 1. PMID 40106374
- See also: D5242C00001_CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5242C00001&attachmentIdentifier=eef527b8-b359-440a-914a-8fc0c1368a17&fileName=D5242C00001_CSP_redacted.pdf&versionIdentifier=
- See also: D5242C00001_SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5242C00001&attachmentIdentifier=735646be-fb1f-4305-9005-ae61b567e45b&fileName=D5242C00001_SAP_redacted.pdf&versionIdentifier=
- See also: D5242C00001_CSR Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5242C00001&attachmentIdentifier=b2542007-d51d-4cfa-9c07-24b5baef06aa&fileName=D5242c00001_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 416 participants were randomized, 6 of which were removed from analyses due to GCP issues, before study unblinding. The remaining 410 were randomized to either the treatment arm (204 participants) or placebo (206 participants) arms of the double-blind treatment period. Two participants were randomized but not dosed (one was withdrawal by subject, one did not meet inclusion/exclusion criteria). Therefore, 203 participants started in the treatment arm and 205 in the placebo arm.
Pre-assignment Details: All patients completed a 5-week run-in period during which inclusion/exclusion criteria were assessed, medical history was recorded, nasal endoscopy and biopsy and CT scan were performed, and patient-reported outcomes (PROs) and clinical laboratory tests were performed.
Groups:
- Tezepelumab: 210 mg tezepelumab injection delivered subcutaneously every 4 weeks + background mometasone furoate (MFNS) or equivalent intranasal corticosteroid (INCS).
- Placebo: Matching Placebo injection delivered subcutaneously every 4 weeks + background mometasone furoate (MFNS) or equivalent intranasal corticosteroid (INCS)
Period: Overall Study
Arm/Group | Tezepelumab | Placebo
Started | 203 | 205
Completed | 193 | 174
Not Completed | 10 | 31
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 8 | 23
Not completed — Severe incompliance | 0 | 1
Not completed — Nasal polyp surgery | 0 | 2
Not completed — Other biologic treatment | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received any IP were included in the full analysis set.
Groups:
- Tezepelumab: 210 mg tezepelumab injection delivered subcutaneously every 4 weeks + background MFNS/INCS.
- Placebo: Matching Placebo injection delivered subcutaneously every 4 weeks + background MFNS/INCS.
- Total: Total of all reporting groups
Arm/Group | Tezepelumab | Placebo | Total
Number analyzed (Participants) | 203 | 205 | 408
Age, Categorical [Count of Participants; unit: Participants] — Age group at screening visit
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 174 | 179 | 353
    >=65 years | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at screening visit
  years | 50.1 (13.60) | 49.4 (13.69) | 49.7 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at screening visit
  Participants
    Female | 77 | 65 | 142
    Male | 126 | 140 | 266
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 192 | 194 | 386
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 3 | 3 | 6
  White | 150 | 149 | 299
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 46 | 51 | 97
  Other | 4 | 2 | 6
  Not reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Polyp Score at Week 52
Description: The total nasal polyp score (NPS) is the sum of the right and left nostril scores (maximum of 8), as evaluated by nasal endoscopy. Higher scores indicate greater symptom severity. The left and right score will be based on a central read with a scale from 0 to 4. Each nasal endoscopy is evaluated by two independent physician reviewers.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -2.458 [-2.681 to -2.234] | -0.380 [-0.611 to -0.148]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in NPS at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — For participants whose NPS data collected after NP surgery were replaced with the worst possible score (WPS). Data collected after SCS for NP were replaced with the worst post-baseline observation prior to the SCS for NP (WOCF). Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p < .0001, ANCOVA — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; Model: Change from baseline in NPS = Treatment + Baseline co-morbid asthma/AERD/NSAID-ERD + Prior NP surgery + Region + Baseline NPS; Difference in Least Squares Means = -2.078, 95% CI 2-sided [-2.399 to -1.757]

2. Primary Outcome: Change From Baseline in Bi-weekly Mean Nasal Congestion Score (NCS) at Week 52
Description: The NCS is captured by one item in the NPSD (nasal polyps symptom diary) asking participants to rate the severity of their worst NC over the past 24 hours using the following response options: 0 - None; 1 - Mild; 2 - Moderate; 3 - Severe. Baseline will be the mean of daily responses from Day -13 to Day 0. Bi-weekly (14-day) mean NCS will be calculated if at least 8 days in each 14-day period has evaluable data; otherwise the bi-weekly mean is set to missing.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -1.743 [-1.864 to -1.622] | -0.703 [-0.830 to -0.577]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in bi-weekly mean NCS at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — For participants whose NCS data collected after NP surgery were replaced with the worst possible score (WPS). Data collected after SCS for NP were replaced with the worst post-baseline observation prior to the SCS for NP (WOCF). Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p < .0001, ANCOVA — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; Model: Change from baseline in bi-weekly mean NCS = Treatment + Baseline co-morbid asthma/AERD/NSAID-ERD + Prior NP surgery + Region + Baseline NCS; Difference in Least Squares Means = -1.039, 95% CI 2-sided [-1.214 to -0.865]

3. Secondary Outcome: Change From Baseline in Bi-weekly Mean Loss of Smell at Week 52
Description: Participant reported sense of smell will be evaluated as part of the NPSD. Loss of smell is captured by the DSS item (difficulty with sense of smell) in the NPSD asking participants to rate the severity of their worst difficulty with sense of smell over the past 24 hours using the following response options: 0 - None; 1 - Mild; 2 - Moderate; 3 - Severe. Baseline will be the mean of daily responses to the from Day -13 to Day 0. Bi-weekly (14-day) mean loss of smell will be calculated if at least 8 days in each 14-day period has evaluable data; otherwise the bi-weekly mean is set to missing.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -1.261 [-1.382 to -1.139] | -0.255 [-0.378 to -0.133]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in bi-weekly mean loss of smell at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — For participants whose loss of smell data collected after NP surgery were replaced with the worst possible score (WPS). Data collected after SCS for NP were replaced with the worst post-baseline observation prior to the SCS for NP (WOCF). Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p < .0001, ANCOVA — The p-value is unadjusted, and is statistically significant at 0.01 level under multiple testing strategy; Change from baseline in bi-weekly mean loss of smell=Treatment+Baseline co-morbid asthma/AERD/NSAID-ERD+Prior NP surgery+Region+Baseline loss of smell; Difference in Least Squares Means = -1.005, 95% CI 2-sided [-1.177 to -0.834]

4. Secondary Outcome: Change From Baseline in SinoNasal Outcome Test 22 (SNOT-22) at Week 52
Description: SinoNasal Outcome Test 22 scores are participant-reported and assess physical problems, functional limitations and emotional consequences of SinoNasal conditions. Patient-reported symptom severity and symptom impact over the past 2 weeks are captured via a 6-point scale (0-No Problem to 5-Problem as bad as it can be). The total score is the sum of item scores and has a range from 0 to 110 (higher scores indicate poorer outcomes).
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -45.022 [-48.572 to -41.472] | -17.580 [-21.189 to -13.971]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in SNOT-22 at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — For participants whose SNOT-22 total score collected after NP surgery were replaced with the worst possible score (WPS). Data collected after SCS for NP were replaced with the worst post-baseline observation prior to the SCS for NP (WOCF). Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p < .0001, ANCOVA — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; Change from baseline in SNOT-22 = Treatment + Baseline co-morbid asthma/AERD/NSAID-ERD + Prior NP surgery + Region + Baseline SNOT-22 total score; Difference in Least Squares Means = -27.441, 95% CI 2-sided [-32.512 to -22.370]

5. Secondary Outcome: Change From Baseline in Lund Mackay Score Evaluated by CT at Week 52.
Description: The Lund-Mackay score scoring system is used to provide a quantitative assessment of nasal sinuses on sinus CT scans. Based on the sinus CT images, the five sinuses (maxillary, anterior ethmoid, posterior ethmoid, sphenoid and frontal) on each site are score by central radiologist as follows: (0-Normal; 1-Partial Opacification; 2-Total Opacification). The osteomeatal complex is scored for right and left sides (0 - Not occluded; 2- Occluded). The total score ranges from 0 to 24 (higher scores indicate poorer outcomes).
Time Frame: Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -6.270 [-6.740 to -5.799] | -0.569 [-1.046 to -0.093]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in LMK at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — For participants whose LMK score collected after NP surgery were replaced with the worst possible score (WPS). Data collected after SCS for NP were replaced with the worst post-baseline observation prior to the SCS for NP (WOCF). Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p < .0001, ANCOVA — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; Change from baseline in LMK score = Treatment + Baseline co-morbid asthma/AERD/NSAID-ERD + Prior NP surgery + Region + Baseline LMK score; Difference in Least Squares Means = -5.700, 95% CI 2-sided [-6.371 to -5.030]

6. Secondary Outcome: Percentage of Participants With Nasal Polyp Surgery Decision and/or Systemic Corticosteroid for Nasal Polyposis up to Week 52
Description: Surgery is defined as any procedure involving instruments resulting in incision and removal of tissue (e.g., polypectomy, endoscopic sinus surgery). Rescue treatment of NP is defined as requiring treatment with systemic corticosteroids (SCS) for at least 3 consecutive days (a single depo-injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids).
  Time to first NP surgery decision or SCS for NP = (date of the first NP surgery decision or start date of first SCS for NP use - date of randomisation)+1.
  Kaplan Meier estimates of percentage of participants with events and 95% confidence interval are provided for each treatment group.
Time Frame: Up to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Percentage of participants | 5.7 [1.3 to 15.0] | 31.4 [25.0 to 38.0]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Hazard ratio of time to first SCS for NP and/or surgery decision (tezepelumab/placebo) = 1; Test type: Superiority; p < .0001, Regression, Cox — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; The Cox regression was adjusted for treatment, baseline co-morbid asthma/AERD/NSAID-ERD status, prior NP surgery status, and region; Hazard Ratio (HR) = 0.08, 95% CI 2-sided [0.03 to 0.16] — A hazard ratio less than 1 indicates a lower rate of incidence for subjects on Tezepelumab

7. Secondary Outcome: Percentage of Participants With Nasal Polyp Surgery Decision up to Week 52
Description: Surgery is defined as any procedure involving instruments resulting in incision and removal of tissue (e.g., polypectomy, endoscopic sinus surgery).
  Time to first NP surgery decision = (date of the first NP surgery decision - date of randomisation)+1.
  Kaplan Meier estimates of percentage of participants with events and 95% confidence interval are provided for each treatment group.
Time Frame: Up to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Percentage of participants | 0.5 [0.0 to 2.5] | 22.0 [16.4 to 28.2]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Hazard ratio of time to first surgery decision (tezepelumab/placebo) = 1; Test type: Superiority; p < .0001, Regression, Cox — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; The Cox regression adjusted for treatment, baseline co-morbid asthma/AERD/NSAID-ERD status, prior NP surgery status, and region; Hazard Ratio (HR) = 0.02, 95% CI 2-sided [0.00 to 0.09] — A hazard ratio less than 1 indicates a lower rate of incidence for subjects on Tezepelumab

8. Secondary Outcome: Percentage of Participants With Systemic Corticosteroids for Nasal Polyposis up to Week 52
Description: Systemic corticosteroids (SCS) for nasal polyposis (NP) is defined as requiring at least 3 consecutive days (a single depo-injectable dose of corticosteroids was considered equivalent to a 3-day course of SCS) for NP.
  Time to first SCS for NP = (start date of first SCS for NP use - date of randomisation)+1.
  Kaplan Meier estimates of percentage of participants with events and 95% confidence interval are provided for each treatment group.
Time Frame: Up to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Percentage of participants | 5.2 [1.1 to 14.7] | 19.3 [14.1 to 25.1]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Hazard ratio of time to first SCS use for NP (tezepelumab/placebo) = 1; Test type: Superiority; p < .0001, Regression, Cox — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.11, 95% CI 2-sided [0.04 to 0.25] — A hazard ratio less than 1 indicates a lower rate of incidence for subjects on Tezepelumab

9. Secondary Outcome: Change From Baseline in Bi-weekly Mean Nasal Polyposis Symptom Diary Total Symptom Score at Week 52
Description: The participant completed the nasal polyposis symptom diary each morning throughout the study. The participant was asked to consider their experience with nasal polyposis/nasal polyps over the past 24 hours when responding to each question. Participants were asked to report their experience with nasal polyposis symptoms (nasal blockage, nasal congestion, runny nose, postnasal drip (mucus drainage down the throat), headache, facial pain, facial pressure, difficulty with sense of smell). Participants reported the severity of each symptom and symptom impact at its worst using a 4-point verbal rating scale (0-None to 3-Severe). A total symptom score (range from 0 to 24) was calculated by taking the sum of the 8 equally weighted symptom items. Higher scores indicate greater symptom severity.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -10.388 [-11.174 to -9.601] | -3.429 [-4.241 to -2.617]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in bi-weekly mean NPSD TSS at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — For participants whose bi-weekly mean NPSD TSS collected after NP surgery were replaced with the worst possible score (WPS). Data collected after SCS for NP were replaced with the worst post-baseline observation prior to the SCS for NP (WOCF). Missing data not due to intercurrent events were imputed using MI (MAR). Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p < .0001, ANCOVA — The p-value is unadjusted and it is statistically significant at 0.01 level under multiple testing strategy; Model: Change from baseline in NPSD TSS = Treatment + Baseline co-morbid asthma/AERD/NSAID-ERD + Prior NP surgery + Region + Baseline NPSD TSS; Difference in Least Squares Means = -6.959, 95% CI 2-sided [-8.085 to -5.833]

10. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume (L) in 1 Second at Week 52.
Description: For participants with comorbid asthma and aspirin exacerbated respiratory disease (AERD)/nonsteroidal anti-inflammatory drug exacerbated respiratory disease (NSAID-ERD), difference in change from baseline in pre-bronchodilator forced expiratory volume in 1 second (FEV1) in the tezepelumab arm as compared to placebo at Week 52. FEV1 is defined as the volume of air exhaled from the lungs in the first second of forced expiration.
Time Frame: Baseline to Week 52
Population: co-morbid asthma/AERD/NSAID-ERD subset (All randomized participants who baseline co-morbid asthma/AERD/NSAID-ERD=Yes).
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 122 | 126
Liter | 0.022 [-0.065 to 0.108] | 0.027 [-0.055 to 0.108]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Null Hypothesis: Difference in mean change from baseline in pre-BD FEV1 at 52 weeks (tezepelumab minus placebo) = 0; Test type: Superiority — Observed pre-BD FEV1 data were used in the analysis regardless of NP surgery and SCS/biologic for NP. Missing data were imputed assuming MAR. Analysis was repeated on 100 imputed datasets, and results were combined using Rubin's formula; p = 0.9362, ANCOVA — The p-value is unadjusted; Model: Change from baseline in pre-BD FEV1 = Treatment + Baseline co-morbid asthma/AERD/NSAID-ERD + Prior NP surgery + Region + Baseline pre-BD FEV1; Difference in Least Squares Means = -0.005, 95% CI 2-sided [-0.121 to 0.111]

11. Other Pre Specified Outcome: Change From Baseline Over Time in Nasal Polyp Score Through Week 52.
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score
  Week 4 | -1.615 [-1.797 to -1.433] | -0.255 [-0.434 to -0.077]
  Week 12 | -1.918 [-2.112 to -1.723] | -0.376 [-0.569 to -0.182]
  Week 24 | -2.104 [-2.310 to -1.899] | -0.314 [-0.522 to -0.106]
  Week 36 | -2.351 [-2.552 to -2.149] | -0.287 [-0.493 to -0.082]
  Week 52 | -2.458 [-2.681 to -2.234] | -0.380 [-0.611 to -0.148]

12. Other Pre Specified Outcome: Proportion of Participants With ≥1 Point Reduction in the Nasal Polyp Score at Week 52
Description: The Nasal Polyp Score is the sum of the right and left nostril scores (maximum 8), as evaluated by nasal endoscopy. A participant with ≥1 point reduction in NPS at Week 52 in the absence of SCS for NP, biologic for NP, or NP surgery at or prior to that time point was defined as a responder, otherwise the participant was defined as a non-responder.
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Participants | 161 | 64

13. Other Pre Specified Outcome: Proportion of Participants With ≥2 Point Reduction in the Nasal Polyp Score at Week 52
Description: The Nasal Polyp Score is the sum of the right and left nostril scores (maximum 8), as evaluated by nasal endoscopy. A participant with ≥2 point reduction in NPS at Week 52 in the absence of SCS for NP, biologic for NP, or NP surgery at or prior to that time point was defined as a responder, otherwise the participant was defined as a non-responder.
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Participants | 129 | 39

14. Other Pre Specified Outcome: Change From Baseline Over Time in Bi-weekly Mean Nasal Congestion Score Evaluated by Nasal Polyposis Symptom Diary Through Week 52.
Description: as for outcome 2
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score
  Week 2 | -0.379 [-0.438 to -0.319] | -0.192 [-0.251 to -0.133]
  Week 4 | -0.779 [-0.868 to -0.691] | -0.322 [-0.411 to -0.234]
  Week 8 | -1.134 [-1.236 to -1.032] | -0.451 [-0.553 to -0.349]
  Week 12 | -1.270 [-1.376 to -1.164] | -0.607 [-0.714 to -0.500]
  Week 24 | -1.515 [-1.628 to -1.402] | -0.703 [-0.818 to -0.588]
  Week 36 | -1.629 [-1.748 to -1.509] | -0.726 [-0.850 to -0.601]
  Week 48 | -1.735 [-1.856 to -1.613] | -0.721 [-0.847 to -0.594]
  Week 52 | -1.743 [-1.864 to -1.622] | -0.703 [-0.830 to -0.577]

15. Other Pre Specified Outcome: Change From Baseline in Loss of Smell Evaluated by University of Pennsylvania Smell Identification Test (UPSIT) at Week 52.
Description: The University of Pennsylvania Smell Identification Test is a quantitative test of olfactory function which uses microencapsulated odorants that are released by scratching standardized odour-impregnated test booklets. Scores are based on number of correctly identified odours (score range 0-40, lower scores indicate poorer outcomes).
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | 9.310 [8.147 to 10.474] | -0.192 [-1.378 to 0.993]

16. Other Pre Specified Outcome: Change From Baseline in Modified Lund Mackay Score Evaluated by CT at Week 52.
Description: The Modified Lund-Mackay score scoring system was used to provide a semi-quantitative assessment of nasal sinuses on sinus CT scans. Based on the sinus CT images, the five sinuses (maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) on each side were scored. Each sinus on each side was scored based on the percentage of opacification from mucosal thickening according to matrix: (score 0 for 0% Opacification; score 1 for 1-25% Opacification; score 2 for 26-50% Opacification; score 3 for 51-75% Opacification; score 4 for 76-99% Opacification; score 5 for 100% Opacification). The range of total Modified Lund Mackay score is from 0 to 50. Higher scores indicate greater symptom severity.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -17.520 [-18.708 to -16.332] | -1.106 [-2.291 to 0.078]

17. Other Pre Specified Outcome: Change From Baseline in Sinus Severity Score by Quantitative CT Assessment at Week 52
Description: Quantitative assessment of sinus CT image data were used to derive an objective measure of sinus disease burden called sinus severity score. The sinus severity score is defined as: (sinus mucosal volume)/(sinus mucosal volume + sinus air volume)×100%. The range of sinus severity score is 0 to 100. Higher scores indicate greater symptom severity.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score | -32.754 [-35.047 to -30.461] | -1.978 [-4.267 to 0.310]

18. Other Pre Specified Outcome: Exposure of Systemic Corticosteroids Over 52 Weeks
Description: The number of courses of SCS for NP per year was analysed using a negative binomial model. The response variable was the number of courses of SCS for NP received by a participant over the planned treatment period.
  The model included treatment group, baseline co-morbid asthma/AERD/NSAID-ERD status, prior NP surgery status, and region as factors. The logarithm of the time at risk (in years) was used as an offset variable, to adjust different follow-up times. Time during a course was not included in the calculation of time at risk.
Time Frame: Over 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: SCS courses per year
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
SCS courses per year | 0.04 [0.02 to 0.08] | 0.35 [0.23 to 0.55]

19. Other Pre Specified Outcome: Change From Baseline by Domain of the Nasal Polyposis Symptom Diary Through Week 52
Description: The participant will complete an 11-item nasal polyposis symptom diary each morning throughout the screening, treatment and follow-up periods. The participant is asked to consider their experience with nasal polyposis/nasal polyps over the past 24 hours when responding to each question. Participants are asked to report their experience with nasal polyposis symptoms (nasal blockage, nasal congestion, runny nose, postnasal drip (mucus drainage down the throat), headache, facial pain, facial pressure, and difficulty with sense of smell) and symptom impacts (difficulty with sleeping due to nasal symptoms and difficulty with daily activities due to nasal symptoms). Participants report the severity of each symptom and symptom impact at its worst using a 4-point verbal rating scale (0-None to 3-Severe).
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Score
  Nasal Blockage Week 2 | -0.359 [-0.416 to -0.301] | -0.170 [-0.227 to -0.112]
  Nasal Blockage Week 4 | -0.744 [-0.831 to -0.656] | -0.298 [-0.385 to -0.211]
  Nasal Blockage Week 8 | -1.122 [-1.225 to -1.018] | -0.423 [-0.527 to -0.320]
  Nasal Blockage Week 12 | -1.259 [-1.367 to -1.152] | -0.555 [-0.663 to -0.447]
  Nasal Blockage Week 24 | -1.502 [-1.617 to -1.387] | -0.678 [-0.795 to -0.561]
  Nasal Blockage Week 36 | -1.628 [-1.750 to -1.506] | -0.703 [-0.830 to -0.576]
  Nasal Blockage Week 48 | -1.697 [-1.821 to -1.573] | -0.722 [-0.850 to -0.594]
  Nasal Blockage Week 52 | -1.759 [-1.882 to -1.636] | -0.697 [-0.825 to -0.569]
  Nasal Congestion Week 2 | -0.379 [-0.438 to -0.319] | -0.192 [-0.251 to -0.133]
  Nasal Congestion Week 4 | -0.779 [-0.868 to -0.691] | -0.322 [-0.411 to -0.234]
  Nasal Congestion Week 8 | -1.134 [-1.236 to -1.032] | -0.451 [-0.553 to -0.349]
  Nasal Congestion Week 12 | -1.270 [-1.376 to -1.164] | -0.607 [-0.714 to -0.500]
  Nasal Congestion Week 24 | -1.515 [-1.628 to -1.402] | -0.703 [-0.818 to -0.588]
  Nasal Congestion Week 36 | -1.629 [-1.748 to -1.509] | -0.726 [-0.850 to -0.601]
  Nasal Congestion Week 48 | -1.735 [-1.856 to -1.613] | -0.721 [-0.847 to -0.594]
  Nasal Congestion Week 52 | -1.743 [-1.864 to -1.622] | -0.703 [-0.830 to -0.577]
  Runny Nose Week 2 | -0.347 [-0.407 to -0.288] | -0.164 [-0.224 to -0.105]
  Runny Nose Week 4 | -0.676 [-0.757 to -0.595] | -0.239 [-0.320 to -0.158]
  Runny Nose Week 8 | -0.966 [-1.056 to -0.875] | -0.360 [-0.450 to -0.270]
  Runny Nose Week 12 | -1.075 [-1.173 to -0.976] | -0.467 [-0.566 to -0.369]
  Runny Nose Week 24 | -1.258 [-1.363 to -1.153] | -0.464 [-0.571 to -0.358]
  Runny Nose Week 36 | -1.353 [-1.466 to -1.240] | -0.467 [-0.583 to -0.351]
  Runny Nose Week 48 | -1.448 [-1.561 to -1.336] | -0.410 [-0.528 to -0.292]
  Runny Nose Week 52 | -1.429 [-1.545 to -1.313] | -0.400 [-0.523 to -0.277]
  Postnasal Drip Week 2 | -0.252 [-0.310 to -0.195] | -0.153 [-0.210 to -0.096]
  Postnasal Drip Week 4 | -0.552 [-0.633 to -0.472] | -0.230 [-0.310 to -0.150]
  Postnasal Drip Week 8 | -0.806 [-0.898 to -0.715] | -0.336 [-0.428 to -0.244]
  Postnasal Drip Week 12 | -0.916 [-1.015 to -0.816] | -0.388 [-0.488 to -0.288]
  Postnasal Drip Week 24 | -1.084 [-1.194 to -0.974] | -0.418 [-0.529 to -0.306]
  Postnasal Drip Week 36 | -1.175 [-1.290 to -1.061] | -0.441 [-0.559 to -0.322]
  Postnasal Drip Week 48 | -1.189 [-1.307 to -1.071] | -0.376 [-0.498 to -0.253]
  Postnasal Drip Week 52 | -1.177 [-1.294 to -1.060] | -0.348 [-0.471 to -0.225]
  Headache Week 2 | -0.259 [-0.318 to -0.199] | -0.185 [-0.245 to -0.126]
  Headache Week 4 | -0.414 [-0.489 to -0.340] | -0.294 [-0.369 to -0.220]
  Headache Week 8 | -0.673 [-0.753 to -0.594] | -0.382 [-0.461 to -0.303]
  Headache Week 12 | -0.753 [-0.842 to -0.665] | -0.439 [-0.528 to -0.350]
  Headache Week 24 | -0.870 [-0.970 to -0.771] | -0.470 [-0.571 to -0.369]
  Headache Week 36 | -0.928 [-1.034 to -0.821] | -0.387 [-0.496 to -0.278]
  Headache Week 48 | -0.962 [-1.075 to -0.849] | -0.361 [-0.476 to -0.245]
  Headache Week 52 | -0.941 [-1.056 to -0.825] | -0.341 [-0.459 to -0.222]
  Facial Pain Week 2 | -0.250 [-0.310 to -0.190] | -0.171 [-0.231 to -0.111]
  Facial Pain Week 4 | -0.438 [-0.514 to -0.363] | -0.276 [-0.352 to -0.201]
  Facial Pain Week 8 | -0.723 [-0.806 to -0.640] | -0.368 [-0.450 to -0.285]
  Facial Pain Week 12 | -0.801 [-0.888 to -0.713] | -0.438 [-0.526 to -0.350]
  Facial Pain Week 24 | -0.957 [-1.056 to -0.858] | -0.494 [-0.594 to -0.393]
  Facial Pain Week 36 | -1.000 [-1.106 to -0.893] | -0.396 [-0.506 to -0.286]
  Facial Pain Week 48 | -1.010 [-1.125 to -0.895] | -0.358 [-0.476 to -0.239]
  Facial Pain Week 52 | -1.002 [-1.118 to -0.886] | -0.316 [-0.436 to -0.197]
  Facial Pressure Week 2 | -0.276 [-0.338 to -0.215] | -0.170 [-0.232 to -0.109]
  Facial Pressure Week 4 | -0.509 [-0.587 to -0.431] | -0.277 [-0.355 to -0.199]
  Facial Pressure Week 8 | -0.778 [-0.866 to -0.689] | -0.373 [-0.461 to -0.284]
  Facial Pressure Week 12 | -0.840 [-0.929 to -0.750] | -0.460 [-0.549 to -0.370]
  Facial Pressure Week 24 | -0.987 [-1.087 to -0.887] | -0.501 [-0.603 to -0.400]
  Facial Pressure Week 36 | -1.039 [-1.148 to -0.930] | -0.400 [-0.512 to -0.288]
  Facial Pressure Week 48 | -1.093 [-1.210 to -0.975] | -0.379 [-0.499 to -0.258]
  Facial Pressure Week 52 | -1.081 [-1.200 to -0.962] | -0.342 [-0.464 to -0.220]
  Difficulty with Sense of Smell Week 2 | -0.126 [-0.164 to -0.088] | -0.037 [-0.074 to 0.001]
  Difficulty with Sense of Smell Week 4 | -0.416 [-0.483 to -0.348] | -0.053 [-0.120 to 0.014]
  Difficulty with Sense of Smell Week 8 | -0.804 [-0.897 to -0.711] | -0.107 [-0.200 to -0.015]
  Difficulty with Sense of Smell Week 12 | -0.909 [-1.015 to -0.804] | -0.208 [-0.313 to -0.103]
  Difficulty with Sense of Smell Week 24 | -1.078 [-1.195 to -0.961] | -0.275 [-0.392 to -0.158]
  Difficulty with Sense of Smell Week 36 | -1.101 [-1.221 to -0.980] | -0.300 [-0.422 to -0.177]
  Difficulty with Sense of Smell Week 48 | -1.242 [-1.364 to -1.121] | -0.289 [-0.413 to -0.166]
  Difficulty with Sense of Smell Week 52 | -1.261 [-1.382 to -1.139] | -0.255 [-0.378 to -0.133]
  Difficulty with Sleeping Week 2 | -0.340 [-0.399 to -0.281] | -0.188 [-0.247 to -0.129]
  Difficulty with Sleeping Week 4 | -0.655 [-0.738 to -0.572] | -0.284 [-0.367 to -0.202]
  Difficulty with Sleeping Week 8 | -0.994 [-1.084 to -0.904] | -0.454 [-0.544 to -0.364]
  Difficulty with Sleeping Week 12 | -1.081 [-1.177 to -0.984] | -0.495 [-0.591 to -0.398]
  Difficulty with Sleeping Week 24 | -1.262 [-1.365 to -1.159] | -0.516 [-0.621 to -0.411]
  Difficulty with Sleeping Week 36 | -1.307 [-1.420 to -1.194] | -0.520 [-0.637 to -0.403]
  Difficulty with Sleeping Week 48 | -1.307 [-1.427 to -1.188] | -0.469 [-0.595 to -0.342]
  Difficulty with Sleeping Week 52 | -1.317 [-1.436 to -1.197] | -0.454 [-0.580 to -0.327]
  Difficulty with Daily Activities week 2 | -0.282 [-0.340 to -0.225] | -0.183 [-0.240 to -0.126]
  Difficulty with Daily Activities week 4 | -0.504 [-0.582 to -0.425] | -0.294 [-0.372 to -0.216]
  Difficulty with Daily Activities week 8 | -0.836 [-0.926 to -0.747] | -0.408 [-0.497 to -0.319]
  Difficulty with Daily Activities week 12 | -0.948 [-1.043 to -0.853] | -0.469 [-0.564 to -0.374]
  Difficulty with Daily Activities week 24 | -1.135 [-1.242 to -1.028] | -0.520 [-0.628 to -0.412]
  Difficulty with Daily Activities week 36 | -1.201 [-1.316 to -1.085] | -0.509 [-0.629 to -0.389]
  Difficulty with Daily Activities week 48 | -1.213 [-1.334 to -1.091] | -0.440 [-0.568 to -0.313]
  Difficulty with Daily Activities week 52 | -1.212 [-1.334 to -1.090] | -0.414 [-0.542 to -0.285]

20. Other Pre Specified Outcome: Change From Baseline in Nasal Peak Inspiratory Flow Through Week 52.
Description: Nasal peak inspiratory flow evaluation represents a physiologic measure of the air flow through both nasal cavities during forced inspiration expressed in liters per minute.
Time Frame: Baseline to Week 52
Population: Full analysis set (All randomized participants who received at least one dose of IP).
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters per minute.
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 205
Liters per minute.
  Week 12 | 21.860 [10.888 to 32.831] | -1.695 [-12.313 to 8.923]
  Week 24 | 29.437 [17.500 to 41.373] | 6.258 [-5.563 to 18.080]
  Week 36 | 11.228 [0.875 to 21.581] | -4.941 [-15.570 to 5.687]
  Week 52 | 22.551 [11.467 to 33.635] | 0.489 [-10.973 to 11.952]

21. Other Pre Specified Outcome: Change From Baseline in Asthma Control Questionnaire-6 at Week 52.
Description: The Asthma Control Questionnaire is an assessment of asthma symptoms (nighttime waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and short acting beta-agonist use). Participants are asked to recall their level of asthma control during the previous week by responding to one bronchodilator use question and 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled).
Time Frame: Baseline to Week 52
Population: Co-morbid asthma/AERD/NSAID-ERD subset
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 122 | 126
Score | -1.203 [-1.334 to -1.072] | -0.815 [-0.967 to -0.663]

22. Other Pre Specified Outcome: Tezepelumab Pharmacokinetics
Description: Serum concentrations of tezepelumab through Week 64. Logarithm transformation was used when calculating geometric mean of serum concentrations. The results were transformed back to original scale.
Time Frame: Pre-dose samples at Baseline, Week 4, Week 12, Week 24, Week 36, Week 52, and Week 64
Population: PK Analysis Set (all participants who received tezepelumab and had at least one detectable tezepelumab serum concentration from a sample collected post-treatment that is assumed not to be affected by factors such as protocol deviations).
  Number analysed at each timepoint is a subset of this based on subjects who had sample results available at that timepoint after analysis window is applied. The placebo arm is not applicable since it is not the experimental product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 203 | 0
μg/mL
  Baseline: number analyzed (Participants) | 189 | 0
  Baseline | NA (NA) — Serum concentrations were not calculable as all 189 participants had concentrations below lower limit of quantification (0.010 μg/mL). |
  Week 4: number analyzed (Participants) | 183 | 0
  Week 4 | 12.165 (35.9) |
  Week 12: number analyzed (Participants) | 175 | 0
  Week 12 | 21.496 (40.8) |
  Week 24: number analyzed (Participants) | 171 | 0
  Week 24 | 23.994 (43.0) |
  Week 36: number analyzed (Participants) | 167 | 0
  Week 36 | 25.237 (45.4) |
  Week 52: number analyzed (Participants) | 167 | 0
  Week 52 | 24.352 (43.7) |
  Week 64: number analyzed (Participants) | 184 | 0
  Week 64 | 2.449 (103.1) |

23. Other Pre Specified Outcome: Immunogenicity of Tezepelumab for Non-China Subjects
Description: Anti-drug antibodies (ADA) responses at baseline and post-baseline. ADA prevalence was defined as patients who are ADA positive at any time including baseline. Persistently positive was defined as having at least two post-baseline ADA positive measurements (with ≥16 weeks between first and last positive) or an ADA positive result at the last available post-baseline assessment. Transiently positive was defined as having at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. Treatment boosted ADA was defined as baseline positive ADA titre that was boosted to a 4-fold or higher-level following treatment. Treatment emergent ADA (ADA incidence) was defined as the sum of treatment induced ADA and treatment boosted ADA.
Time Frame: Pre-dose samples at Baseline to Week 64
Population: Non-China subjects in Safety analysis set (All participants who received at least one dose of IP).
  Number analysed of each ADA category is a subset of this based on subjects who met the definition and had sample results available after analysis window is applied.
Measure: Number; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 174 | 171
Participants
  ADA prevalence | 10 | 19
  ADA positive at baseline only: number analyzed (Participants) | 164 | 162
  ADA positive at baseline only | 2 | 1
  Treatment-induced ADA positive: number analyzed (Participants) | 164 | 162
  Treatment-induced ADA positive | 6 | 12
  Treatment-boosted ADA positive: number analyzed (Participants) | 164 | 162
  Treatment-boosted ADA positive | 0 | 0
  Treatment emergent ADA (ADA incidence): number analyzed (Participants) | 164 | 162
  Treatment emergent ADA (ADA incidence) | 6 | 12
  Both baseline and at least one post-baseline ADA positive: number analyzed (Participants) | 164 | 162
  Both baseline and at least one post-baseline ADA positive | 2 | 4
  ADA persistently positive | 4 | 11
  ADA transiently positive | 4 | 7
  TE-ADA positive with maximum titre > median of maximum titres: number analyzed (Participants) | 164 | 162
  TE-ADA positive with maximum titre > median of maximum titres | 1 | 2
  ADA positive at baseline (regardless of post-baseline): number analyzed (Participants) | 164 | 162
  ADA positive at baseline (regardless of post-baseline) | 4 | 2
  Any post-baseline ADA positive | 8 | 18
  nAb positive at baseline and/or post-baseline (nAb prevalence) | 2 | 2
  Treatment-induced nAb positive (nAb incidence): number analyzed (Participants) | 164 | 162
  Treatment-induced nAb positive (nAb incidence) | 1 | 2

24. Other Pre Specified Outcome: Immunogenicity of Tezepelumab for China Subjects
Description: as for outcome 23
Time Frame: Pre-dose samples at Baseline to Week 64
Population: China subjects in Safety analysis set (All participants who received at least one dose of IP).
  Number analysed of each ADA category is a subset of this based on subjects who met the definition and had sample results available after analysis window is applied.
Measure: Number; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 29 | 34
Participants
  ADA prevalence | 3 | 4
  ADA positive at baseline only: number analyzed (Participants) | 28 | 34
  ADA positive at baseline only | 1 | 0
  Treatment-induced ADA positive: number analyzed (Participants) | 28 | 34
  Treatment-induced ADA positive | 2 | 3
  Treatment-boosted ADA positive: number analyzed (Participants) | 28 | 34
  Treatment-boosted ADA positive | 0 | 0
  Treatment emergent ADA (ADA incidence): number analyzed (Participants) | 28 | 34
  Treatment emergent ADA (ADA incidence) | 2 | 3
  Both baseline and at least one post-baseline ADA positive: number analyzed (Participants) | 28 | 34
  Both baseline and at least one post-baseline ADA positive | 0 | 1
  ADA persistently positive | 1 | 2
  ADA transiently positive | 1 | 2
  TE-ADA positive with maximum titre > median of maximum titres: number analyzed (Participants) | 28 | 34
  TE-ADA positive with maximum titre > median of maximum titres | 1 | 0
  ADA positive at baseline (regardless of post-baseline): number analyzed (Participants) | 28 | 34
  ADA positive at baseline (regardless of post-baseline) | 1 | 1
  Any post-baseline ADA positive | 2 | 4
  nAb positive at baseline and/or post-baseline (nAb prevalence) | 1 | 0
  Treatment-induced nAb positive (nAb incidence): number analyzed (Participants) | 28 | 34
  Treatment-induced nAb positive (nAb incidence) | 1 | 0

ADVERSE EVENTS:
Time Frame: From visit 1 (the date of the first study procedure) until end of study up to week 76.
Description: For analysis of Adverse Events Safety analysis set is used. Safety analysis set : All randomized participants who received at least one dose of study drug.
  AEs occurring during run-in period: date of Visit 1 ≤ AE onset date < date of first dose of IP.
  AEs occurring during on-study period: date of first dose of IP ≤ AE onset date ≤ study completion or withdrawal date.
Groups:
- Run-in Period: Background mometasone furoate (MFNS) or equivalent intranasal corticosteroid (INCS) only.
Arm/Group | Run-in Period | Tezepelumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/408 | 0/203 | 1/205
Serious Adverse Events (participants affected / at risk) | 0/408 | 11/203 | 14/205
Other Adverse Events (participants affected / at risk) | 20/408 | 119/203 | 119/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (N=408) | Tezepelumab (N=203) | Placebo (N=205)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myopericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Graves' disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (N=408) | Tezepelumab (N=203) | Placebo (N=205)
COVID-19 (Infections and infestations) | 1 (1) | 55 (58) | 44 (47)
Nasopharyngitis (Infections and infestations) | 4 (4) | 45 (63) | 23 (42)
Pharyngitis (Infections and infestations) | 0 (0) | 11 (13) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 23 (26) | 13 (16)
Headache (Nervous system disorders) | 11 (11) | 19 (30) | 16 (22)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 12 (15)
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (26) | 56 (104)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (15) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and/or the Principal Investigator shall not include in or shall remove from any proposed publication any Confidential Information, errors or inaccuracies; and shall withhold publication, submission for publication or presentation for a period of ninety (90) days from the date on which the Company receives the material to allow the Company to take such measures as the Company considers necessary to preserve its proprietary rights and/or protect its Confidential Information.

DOCUMENTS (2):
  • Study Protocol (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04851964/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04851964/SAP_001.pdf